CLINICAL TRIAL: NCT01389661
Title: Regeneration of Maxillary Bone Cystic Cavities by Bio Implant of MSHV-H Cells Associated to a Cross-linked Serum Scaffold
Brief Title: Treatment Of Maxillary Bone Cysts With Autologous Bone Mesenchymal Stem Cells (MSV-H)
Acronym: BIOMAX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Sanidad de Castilla y León (Other); University of Valladolid (Other); Centro en Red de Medicina Regenerativa de Castilla y Leon (Other); Citospin (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TerCel0002; 2010-024246-30 (EudraCT Number); EC10-255 (Other Grant/Funding Number: Spanish Ministry of Health, Programa de Terapias Avanzadas); BIOMAX-VA-2010 (Registry Identifier: Protocol Code)
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Maxillary Cyst; Bone Loss of Substance
Keywords: Maxillary bone cysts; Cell therapy; Mesenchymal stem cells; Autologous serum scaffold

STUDY DESIGN:
Intervention Model Description: MSV-H autologous transplantation: Mesenchymal stem cells from bone marrow expanded by GMP-compliant procedure in IBGM cell production unit in autologous plasma scaffold and implanted in maxillary bone cavities after cyst removal
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSV treatment (Experimental): MSV treatment: Mesenchymal stem cells from bone marrow expanded by GMP-compliant procedure in IBGM cell production unit in autologous plasma scaffold and implanted in maxillary bone cavities after cyst removal
  Interventions: Biological: MSV treatment

INTERVENTIONS:
Biological: MSV treatment — Autologous maxillary bone marrow mesenchymal stem cells (MSV-H) collected from patient, mesenchymal cells isolation and expansion under GMP conditions following the IBGM-Valladolid protocol (MSV)
  Other Names: H-MSV, Human Mesenchymal Stem Cells from Valladolid

SUMMARY:
This trial pretends to validate for clinical use a bioengineered product composed of MSV cells (mesenchymal stem cells produced by IBGM, Valladolid, which have already been approved by the Spanish Regulatory Agency for three previous clinical trials) and a cross-linked matrix of autologous plasma patented by The Blood and Tissue Bank of Asturias (WO2008/ 119855) for bone maxillary cysts refilling. These two groups collaborate in the present project with the team of Maxillofacial Surgery of the Hospital Universitario del Río Hortega, who leads the clinical trial and deals with the medical aspects. The proposed trial is based on positive results obtained in previous animal studies performed by the present multidisciplinary team. The investigators propose a phase I / II clinical trial with 10 patients suffering from bone cysts in the maxillofacial region. Autologous mesenchymal stem cells isolated from a bone marrow sample will be seeded in the autologous plasma matrix and cultivated for 3 weeks. At this time, the cyst will be removed by surgery and the cavity filled with the protein matrix containing the mesenchymal cells. Checks will be conducted at 3 weeks, 3 and 6 months following the evolution of the cavity by panoramic radiography and computerized tomography scan.

DETAILED DESCRIPTION:
The objective of this project is to provide a competitive clinical solution with an autologous product, a balanced cost and the possibility of extending use to other pathologies.

This protocol includes treatment of 10 patients with cystic disease of the jaws that meet all the inclusion criteria and none of the exclusion criteria.

For autologous cell preparation a sample of spongy bone from the maxillary tuberosity and 20 ml of serum are obtained from the patient in order to prepare the crosslinked protein matrix and the MSV-H cells. Cells are selected and expanded under GMP conditions according to the methodology used in previous trials (EudraCT 2005-005498-36, 2008-001191-68 and 2009-0170450-11 ). MSV-H cells are obtained directly from biopsy culture jawbone of the patient by cultivation techniques "in vitro" and differentiate for 21 days once conveyed in the matrix with osteogenic differentiation medium of the following composition: DMEM, 10% FBS, 1% P / E, 0.1 mM dexamethasone, 50 mM ascorbate 2-phosphate, 10 mM phosphate ßGlicerol. All differentiation factors have already been approved for clinical use. After the period of the product differentiation can be implanted to the patient.

The bioimplant is used to refill the bone defects after osteotomy and maxillary cyst enucleation, with 5-10 million cells per unit of 2 cm in diameter and 0.3 cm thick. The cavity is closed with the mucoperiosteal flap and sutured with reabsorbable material. The end point of the trial is to evaluate the feasibility, safety and indications of treatment efficacy according to both clinical criteria and objective imaging confirming the volumetric bone regeneration and maintenance over time. For this purposes orthopantomography exploration will be performed before and 2 and 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Maxillar bone cyst with diameter larger than 2 cm and smaller than 4 cm
* Understanding and written acceptance of assay conditions
* Informed written consent of the patient for assay and for surgery
* In women, negative pregnancy test at t=0
* In women, compromise of using anticonceptive methods during the study

Exclusion Criteria:

* Age under 18 or over 65
* Incapacity or legal dependence
* Pregnancy, lactancy, or enrollment in fertility programs
* Previous or concomitant oncological processes.
* Positive serology for HIV-1 orHIV-2, Hepatitis B (HBsAg, Anti-HCV-Ab) or Hepatitis C (Anti-HCV-Ab).
* Immunocompromised patients
* Systemic disease with potential effects on bone metabolism
* Congenital or acquired maxillofacial malformation
* Patients with prescription of drugs acting on bone metabolism, suc as glucocorticoids and bisphosphonates
* Active or recent infection of the cyst
* Recidive of the cyst (previous surgery)
* Participation in other trials or studies in the last 3 months.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and safety of the implementation of MSV in the treatment of maxillary cysts | up to 6 months
  Clinical review and orthopantomograpy at different periods (0, 2 weeks, 2 months and 6 months) assessing evolution from baseline and possible complications.

SECONDARY OUTCOMES:
Indication of efficacy | up to 6 months
  Imaging exploration to evaluate effectiveness through development of criteria for orthopantomography and bone-CT quantitative bone regeneration Evolution at 2 and 6 months from intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Redondo, MD, PhD, Principal Investigator — Oral and Maxillofacial Surgeon, Río Hortega University Hospital, SACYL, Valladolid, Spain; Ana Sánchez, MD, PhD, Study Director — Instituto de Biología y Genética Molecular (IBGM), University of Valladolid, Spain; Javier García-Sancho, MD, PhD, Study Director — University of Valladolid, Spain; Jose Becerra, PhD, Study Director — Centro Andaluz de Nanomedicina y Biotecnología (BIONAND), Universidad de Málaga, Ciber-bbn. Málaga, Spain.
Locations (3):
- Spain (3):
  - Río Hortega University Hospital, Valladolid, Valladid
  - Bionand, Parque Tecnológico de Andalucía, Universidad de Málaga, Málaga
  - Instituto de Biologia y Genetica Molecular, Valladolid

REFERENCES:
- [Derived] Redondo LM, Garcia V, Peral B, Verrier A, Becerra J, Sanchez A, Garcia-Sancho J. Repair of maxillary cystic bone defects with mesenchymal stem cells seeded on a cross-linked serum scaffold. J Craniomaxillofac Surg. 2018 Feb;46(2):222-229. doi: 10.1016/j.jcms.2017.11.004. Epub 2017 Nov 16. PMID 29229365
- See also: Spanish Cell Therapy Network — http://red-tercel.com
- See also: Cell production, Instituto de Biologia y Genetica Molecular (IBGM) University of Valladolid — http://www.ibgm.med.uva.es
- See also: Diseases, Jaw; Jaw Disease — http://www.ncbi.nlm.nih.gov/mesh/68007571